CLINICAL TRIAL: NCT03237637
Title: Comparative Study to Evaluate the Effectiveness of Atenolol and Propranolol in the Treatment of Infantile Hemangiomas
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Raihan Ashraf, Junior Resident, Department of Dermatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INT/IEC/2017/322
Record Dates: First submitted 2017-07-18; First posted 2017-08-02 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Infantile Hemangioma
MeSH Terms: conditions — Hemangioma, Capillary | interventions — Propranolol; Atenolol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A- Propranolol (Active Comparator): Oral propranolol 1mg/kg/day as crushed tablets, in two divided doses, increased to 2mg/kg/day in two divided doses after 24 hours if tolerated well. Treatment will be stopped at complete clinical clearance of lesion (defined arbitrarily as >90% reduction in the size of Infantile Hemangioma as assessed by Physician Global Assessment) or after 9 months of treatment (primary end point) whichever is earlier.
  Interventions: Drug: oral propranolol
- Group B- Atenolol (Experimental): Oral atenolol 0.5mg/kg as a single dose, increased to 1mg/kg as a single dose after 24 hours if tolerated well. Treatment will be stopped at complete clinical clearance of lesion (defined arbitrarily as >90% reduction in the size of Infantile Hemangioma as assessed by Physician Global Assessment) or after 9 months of treatment (primary end point) whichever is earlier.
  Interventions: Drug: oral atenolol

INTERVENTIONS:
Drug: oral propranolol — oral propranolol 1-2mg/kg/day as crushed tablets in two divided doses
  Arms: Group A- Propranolol
Drug: oral atenolol — oral atenolol 0.5-1mg/kg/day as crushed tablets in a single dose
  Arms: Group B- Atenolol

SUMMARY:
Through this study, the investigators shall compare the effectiveness of atenolol with propranolol in the treatment of IH. In addition, the investigators shall try to elucidate the mechanism of action of beta blockers by assessing their action on triggers such as hypoxia. The study design will be a parallel group comparative study wherein patients of IH will be randomized into two groups. One group will receive propranolol and the other atenolol for a maximum period of 9 months. The patients will then be followed up regularly for regression of the IH based on Physician global assessment, hemangioma activity score(HAS), serial photography and lesional ultrasonography. Any side effects encountered during the treatment period will also be noted. Also serial measurements of hypoxia inducible factor 1 alpha(HIF-1α) will be made to ascertain the mechanism of action of the drugs.

DETAILED DESCRIPTION:
AIMS AND OBJECTIVES:

1. To compare the effectiveness and safety of oral atenolol versus oral propranolol in the treatment of infantile hemangiomas.
2. To elucidate the mechanism of action of atenolol and propranolol in the treatment of infantile hemangiomas.

STUDY DESIGN MATERIALS AND METHODS:

This investigator-initiated, prospective, observer blinded, parallel group comparative study on the effect of oral medication in infantile cutaneous hemangiomas is being conducted in the Department of Dermatology, Venereology and Leprology, and Pediatric Surgery, Post Graduate Institute of Medical Education and Research, after getting approval from the institutional Research and Ethics Committee.

Sample size: As this is a pilot study, an arbitrary sample size of 60 (30 in each group) was decided to be kept.

BASELINE CLINICAL ASSESSMENT:

Children satisfying the inclusion and exclusion criteria will be recruited into the study after obtaining an informed consent from the parents. Upon recruitment, each lesion will be evaluated clinically for size, colour, consistency and the phase of evolution- whether proliferative, plateau or regressing. Photographs will be taken along with Physician Global assessment scale and hemangioma activity score (HAS).26 Heart rate, BP, oxygen saturation, ECG , respiratory rate and random blood sugar will be recorded to rule out treatment contraindications. In patients with eyelid involvement, ophthalmologic examinations will be done. These observations will be noted in the case record form.

All patients will be admitted for 48 hours at initiation of treatment and escalation of dosage to record and monitor all parameters- heart rate, BP, blood sugar, oxygen saturation and respiratory rate.

RANDOMISATION, ALLOCATION, CONCEALMENT AND TREATMENT PROTOCOL Upon inclusion, patients will be randomized into two groups; group A and group B, using a computer generated sequence (block randomization). Efforts will be made to reduce recruitment bias by the following allocation concealment. Patients will be screened by Dr Raihan Ashraf and recruited by Dr Sanjeev Handa, Dr Dipankar De and Dr Muneer Abas. Allocation to either group will be done by Mrs Asha based on block randomization. Thereafter, Dr Rahul Mahajan will prescribe the oral drug based on the group to which the patient is allotted such that the parents of the patient are not blinded to the drug administered. The child shall be admitted to Advanced Paediatric Centre for monitoring of parameters by Dr Raihan Ashraf. At follow up assessment will be done by Dr Raihan Ashraf blinded to the randomization and allocation.

Evaluation of improvement will be done by the following means

1. Physician Global Assessment: Score will be calculated by an independent dermatologist blinded to the management protocol with the help of photographs, at baseline and monthly thereafter. Serial Photography will be done at every 4 weeks.

   (The lesion will be photographed with and without flash with a standard 12 pixel digital camera at 30cm distance and approximately 180 dpi resolution)
2. HAS. Score will be calculated at baseline and monthly thereafter.
3. Ultrasonography : to objectively assess the size and depth of hemangioma will be done at baseline, 6 months and 9 months.

RECORDING OF ADVERSE EVENTS:

All the subjects will be reviewed at 1 month intervals. A full clinical examination will be performed during each visit, including growth chart measurements and cardiovascular status and any side effects like sleep disturbances, hypoglycemia, hypotension will be recorded in the case record form. Mild side effects will be recorded and managed. Serious side effects will be reported to the Safety committee and the patient withdrawn from the study.

LABORATORY EVALUATION Serum Hypoxia inducible factor 1α (HIF-1α) will be measured by ELISA at baseline and 9 months or completion of treatment.

PRIMARY OUTCOME MEASURES:

1. Mean difference in

   1. Number of patients achieving complete clinical clearance of lesion (PGA Score of 5) in the two groups
   2. Number of days required to achieve complete clinical clearance of lesion (PGA Score of 5) in the two groups
   3. Mean decrease in the volume of lesions in the two groups
   4. Mean decrease in HAS in the two groups
2. Frequency of adverse effects (minor and serious) in Group A versus Group B.

SECONDARY OUTCOME MEASURES:

1. Mean difference in HIF-1α levels before and after treatment in Group A and Group B.

STATISTICAL ANALYSIS The statistical analysis will be carried out using Statistical package for Social Sciences (SPSS Inc.,Chicago IL, version 15.0 Windows). The analysis will be done both for Per Protocol population( PP) as well as the Intention to Treat( ITT) population as primary population for analysis. All quantitative variables will be estimated using measures of central location (mean, median) and measures of dispersion (standard deviation and standard error). Normality of data will be checked by measures of skewness and Kolmogorov Smirnov tests of normality. For normally distributed data means will be compared using student's t test for groups. For skewed data Mann Whitney test will be applied for group. Qualitative or categorical variables will be described as frequencies and proportions. Proportions will be compared using Chi square or Fischer's exact test whichever is applicable. All statistical tests will be two sided and performed at a significance of α=0.05.

ETHICAL JUSTIFICATION Since the widespread use of propranolol for the use of infantile hemangiomas, there have come to light various side effects it may cause. Though usually mild and few, rare complications like asymptomatic hypoglycemia, hypotension and bronchial hyperreactivity can be life threatening. The proposed study aims to overcome these side effects with the use of cardio selective beta blocker atenolol which have safely been used in infants previously for cardiological indications like arrhythmias. In addition, it gives a reasonable treatment alternative for infants in whom propranolol is contraindicated. Furthermore, the exact magnitude of CNS effects resulting from propranolol use, especially in the early developmental stages is not currently known. Impairment in short- and long-term memory, psychomotor function, sleep quality and mood have been reported. These effects may not be readily recognizable and require specialized assessment of cognitive function not routinely performed. Furthermore, there may be a delay between exposure and cognitive defects. These side effects would theoretically be alleviated with the use of atenolol due to its impermeability through the blood brain barrier.

The investigations planned are necessary for the optimum management of participants. All blood samples will be taken with a 26 gauge needle so that there is minimal pain and discomfort to the patient and the amount of blood drawn for investigations will not cause any haemodynamic instability.

According to the guidelines set up by ICMR (1994) and Helsinki declaration (modified 2000), the following will be adhered in all patients enrolled in the study:

* The patients involved in the research project will be informed participants.
* Each patient will be adequately informed of the aims, methods, the anticipated benefits and potential risks of the study and the discomfort it may entail to him/her and the remedies thereof.
* Every precaution will be taken to respect the privacy of the patient, the confidentiality of the patient's information and to minimize the impact of the study on his/her physical and mental integrity and his/her personality.
* The patient will be given the right to abstain from participation in the study or to withdraw consent to participate at any time of the study without reprisal.
* Due care and caution will be taken at all stages of the research to ensure that the patient is put to the minimum risk, suffer from no irreversible adverse effects and, generally, benefit from and by the research or experiment.
* Written informed consent will be obtained from all the patients included in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Children diagnosed with problematic infantile hemangiomas

   1. Potentially disfiguring infantile hemangiomas at any site.
   2. Functionally threatening infantile hemangiomas near the eyes, nose, natural orifices, limbs, genitalia.
   3. Ulcerated infantile hemangiomas.
   4. Segmental infantile hemangiomas.
   5. Uncomplicated progressive infantile hemangiomas with unpredictable future course.
2. Age group: less than 1 year of age.
3. Either sex
4. Multiple hemangiomas

Exclusion Criteria:

1. Infants with heart disease, cardiac arrhythmias
2. Broncho -obstructive disease.
3. Premature infants with corrected age less than 40 weeks.
4. Known hypoglycemia
5. Diabetes mellitus
6. Hypertension
7. Hypotension
8. Liver failure
9. Visceral hemangiomas
10. PHACES syndrome

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Mean difference in number of patients achieving complete clinical clearance of lesion (PGA Score of 5) in the two groups | 9 months
  Physician Global Assessment
  Responses to therapy (change of thickness, color, and area) will be recorded on each follow up.The therapeutic responses will be evaluated on a score of 1-5 as follows by an independent dermatologist who will not know the therapies:
  Score 5: >90% improvement or complete clinical involution Score 4: excellent improvement(75-90% decrease) Score 3: good improvement(50-74% decrease) Score 2: minimal improvement( 25-49% decrease) Score 1: poor improvement(1-24% decrease) Score 0: failure (no difference or regrowth)
Mean difference in number of days required to achieve complete clinical clearance of lesion (PGA Score of 5) in the two groups | 9 months
Mean difference in Hemangioma Activity Score in the two groups | 9 months
  Hemangioma Activity score
  Patient name:
  Age:
  Location of infantile hemangioma:
  ("Bright red edge" should only be scored when the HOI is not totally "bright red" Skin colored after activity". Do not score in deep HOI (deep swelling) unless the HOI has changed into it after activity)
  Date
  Deep swelling:
  tense HOI(6) 'neutral' HOI at t=0 or less than 50% reduction at follow up(4) >=50% reduction at follow up (2) No more swelling at follow up (0)
  Bright red/ shining red HOI(5) OR bright red edge(4) Matt red/reddish purple HOI/ matt red edge(3) Blue HOI or Blue shining through in deep HOI(2) Grey HOI(1) Skin colored after activity(0)
  Total score:
  Number of items scored Preliminary HAS= total score/number of items scored
  Ulcer=<1cm2 (+0.5) Ulcer 1-25cm2(+1) Ulcer >=25cm2(+2) HAS= preliminary HAS + ulcer score
Frequency of adverse effects (minor and serious) in the two groups | 9 months

SECONDARY OUTCOMES:
Mean difference in HIF-1α levels before and after treatment in Group A and Group B | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No